CLINICAL TRIAL: NCT05669638
Title: A Prospective Study to Observe Adverse Effects in Patients Receiving Anti-PD1 Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: hongyanli1
Record Dates: First submitted 2022-11-21; First posted 2023-01-03 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Immunotherapy; ADR
Keywords: PD1; immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Blood sample of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about in the development process of adverse reactions of anti-PD1 immunotherapy. The main question it aims to observe:

* The autoantibody profile of patients
* The adverse reactions of patients
* The changes of immune cells and cytokine in patients

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the development process of adverse reactions of anti-PD1 immunotherapy. The main question it aims to observe:

* The autoantibody profile of patients
* The adverse reactions of patients
* The changes of immune cells and cytokine in patients (e.g., T cell, B cell, IL-6, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Receiving anti-PD1 immunotherapy

Exclusion Criteria:

1. Vital signs are unstable
2. Functional impairment of immune system caused by other diseases or other reasons, such as Systemic lupus erythematosus (SLE), AIDS, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving anti-PD1 immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Autoantibodies | Day 1
  Including autoantibodies in Autoimmune encephalitis (NMDAR, AMPA1, AMPA2, CASPR2, GABABR, DPPX, IgLON5 and LGI1), myasthenia gravis (Including AChR, MuSK, LRP4, RyR, Titin), paraneoplastic neurologic syndromes (Hu, Yo, Ri, CV2, PNMA2, Amphiphysin, Recoverin, SOX1, Titin, Zic4, GAD65, Tr) and against gangliosides (GM1, GM2, GM3, GM4, GD1a, GD1b, GD2, GD3, GT1a, GT1b, GQ1b, Sulfatides).
  Cell transfection, ELISpot and ELISA are designed to be used.
Autoantibodies | Week 9
  Including autoantibodies in Autoimmune encephalitis (NMDAR, AMPA1, AMPA2, CASPR2, GABABR, DPPX, IgLON5 and LGI1), myasthenia gravis (Including AChR, MuSK, LRP4, RyR, Titin), paraneoplastic neurologic syndromes (Hu, Yo, Ri, CV2, PNMA2, Amphiphysin, Recoverin, SOX1, Titin, Zic4, GAD65, Tr) and against gangliosides (GM1, GM2, GM3, GM4, GD1a, GD1b, GD2, GD3, GT1a, GT1b, GQ1b, Sulfatides).
  Cell transfection, ELISpot and ELISA are designed to be used.
Autoantibodies | Week 21
  Including autoantibodies in Autoimmune encephalitis (NMDAR, AMPA1, AMPA2, CASPR2, GABABR, DPPX, IgLON5 and LGI1), myasthenia gravis (Including AChR, MuSK, LRP4, RyR, Titin), paraneoplastic neurologic syndromes (Hu, Yo, Ri, CV2, PNMA2, Amphiphysin, Recoverin, SOX1, Titin, Zic4, GAD65, Tr) and against gangliosides (GM1, GM2, GM3, GM4, GD1a, GD1b, GD2, GD3, GT1a, GT1b, GQ1b, Sulfatides).
  Cell transfection, ELISpot and ELISA are designed to be used.
Autoantibodies | Week 33
  Including autoantibodies in Autoimmune encephalitis (NMDAR, AMPA1, AMPA2, CASPR2, GABABR, DPPX, IgLON5 and LGI1), myasthenia gravis (Including AChR, MuSK, LRP4, RyR, Titin), paraneoplastic neurologic syndromes (Hu, Yo, Ri, CV2, PNMA2, Amphiphysin, Recoverin, SOX1, Titin, Zic4, GAD65, Tr) and against gangliosides (GM1, GM2, GM3, GM4, GD1a, GD1b, GD2, GD3, GT1a, GT1b, GQ1b, Sulfatides).
  Cell transfection, ELISpot and ELISA are designed to be used.
Autoantibodies | Week 45
  Including autoantibodies in Autoimmune encephalitis (NMDAR, AMPA1, AMPA2, CASPR2, GABABR, DPPX, IgLON5 and LGI1), myasthenia gravis (Including AChR, MuSK, LRP4, RyR, Titin), paraneoplastic neurologic syndromes (Hu, Yo, Ri, CV2, PNMA2, Amphiphysin, Recoverin, SOX1, Titin, Zic4, GAD65, Tr) and against gangliosides (GM1, GM2, GM3, GM4, GD1a, GD1b, GD2, GD3, GT1a, GT1b, GQ1b, Sulfatides).
  Cell transfection, ELISpot and ELISA are designed to be used.
the change of immune-related adverse events | baseline to Week 45
  Including polyradiculopathies, neuropathies, myasthenic syndromes, myopathies, hypophysitis, aseptic meningitis, encephalitis, multiple sclerosis and other complications.

SECONDARY OUTCOMES:
the immune cell (Including T cell, B cell, etc.) | Day 1
  Including T cell, B cell, etc. Using flow cytometry
the immune cell (Including T cell, B cell, etc.) | Week 9
  Using flow cytometry
the immune cell (Including T cell, B cell, etc.) | Week 21
  Using flow cytometry
the immune cell (Including T cell, B cell, etc.) | Week 33
  Using flow cytometry
the immune cell (Including T cell, B cell, etc.) | Week 45
  Using flow cytometry
the cytokine | Day 1
  Including IL-6, IL-17, etc.
the cytokine | Week 9
  Including IL-6, IL-17, etc.
the cytokine | Week 21
  Including IL-6, IL-17, etc.
the cytokine | Week 33
  Including IL-6, IL-17, etc.
the cytokine | Week 45
  Including IL-6, IL-17, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Li, MD,PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China